CLINICAL TRIAL: NCT03101358
Title: Phase 1/2 Dose-Rising, Safety, Tolerability and Efficacy Study of Topical SOR007 for Cutaneous Metastases
Brief Title: Study of Topical SOR007 Ointment for Cutaneous Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SOR007-2017-01
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Cutaneous Metastasis
Keywords: cutaneous metastases; cutaneous metastasis; skin metastases; skin metastasis
MeSH Terms: interventions — Ointments

STUDY DESIGN:
Intervention Model Description: Phase 1/2, open-label, dose-rising trial of three concentrations of SOR007 (0.15%, 1.0%, 2.0%).
  During the dose escalation phase, the study will follow a standard 3+3 dose-ascending design. If a single dose limiting toxicity (DLT) is identified in one of three subjects in the cohort, a further three subjects will be enrolled at the same dose level. If one or more DLT occur in the three additional subjects enrolled in the cohort, dose escalation will stop and the prior dose level will be regarded as the Maximum Tolerated Dose (MTD) and taken forward into the dose expansion phase. If no further DLT are identified, dose escalation will continue, until either a DLT is identified at a higher dose or the top dose of 2% is reached.
  In the dose expansion phase, additional subjects will be enrolled up to a maximum of 12 subjects at the dose determined to be the MTD (or the top dose, 2.0% SOR007).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SOR007 0.15% (Experimental): 0.15% SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment applied topically twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment
- SOR007 1.0% (Experimental): 1.0% SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment applied topically twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment
- SOR007 2.0% (Experimental): 2.0% SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment applied topically twice daily for 28 days or up to 56 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment

INTERVENTIONS:
Drug: SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment — One (1) Finger Tip Unit (FTU), or approximately 0.5 g, of SOR007 ointment will be applied topically to a 50 cm2 treatment area.

SUMMARY:
This study evaluates a topical nanoparticle paclitaxel ointment (SOR007) for the treatment of cutaneous metastases from non-melanoma cancer in adults. Three concentrations of SOR007 will be evaluated in dose-rising cohorts of three. An expanded cohort will treat additional subjects at the maximum tolerated dose.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, dose-rising study evaluating the safety, tolerability and preliminary efficacy of three concentrations of SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment (0.15%, 1.0%, and 2.0%) applied to non-melanoma cutaneous metastases. A treatment area of 50 cm2 will be selected by the Investigator. Using a gloved hand, subjects will apply one Finger Tip Unit (FTU) of SOR007 to the 50 cm2 treatment area twice daily at approximately the same time each day for 28 days, with the option of extending treatment an additional 28 days to total 56 days for subjects in the dose expansion phase. At each visit (Days 1, 8, 15, 29, and 43 for 28 treatment days; Days 8, 15, 29, 57, and 70 for 56 treatment days), at least two global and two close-up color photographs of the treatment area will be taken (with a ruler for scale). The photographs will be analyzed with ImageJ. Eligible lesions will be determined at baseline by the RECIST definition of measurable tumors (≥ 10mm in its longest diameter). The study will include a dose escalation phase and a dose expansion phase.

In the dose escalation phase, formal safety reviews will be conducted after the last subject in each cohort of three subjects completes 15 days of treatment. The next dose level will enroll upon a finding of safety and tolerability. The top dose or the maximum tolerated dose (if DLT occurs) will be taken into the dose expansion phase and additional subjects will be enrolled to reach a maximum of 16 subjects at that dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Male and female patients ≥ 18 years of age;
3. Malignancies resulting in cutaneous metastasis originating from: breast, lung, head and neck, pancreatic, urinary bladder, prostate, testicular, ovarian, uterine, cervical, gastric, adrenal, thyroid, parathyroid cancers, or other solid tumors;
4. Cutaneous metastases diagnosis confirmed prior to consent by preferred institutional methodology which may include, but is not limited to: biopsy; conventional radiography; imaging techniques to include bone scan (scintigraphy), computed tomography (CT), fluorodeoxyglucose-positron emission tomography (FDG-PET)/CT), magnetic resonance imaging (MRI), F-fluoromisonidazole-(F-FMISO) PET/CT, fluorothymidine-(FLT) PET/CT, fluoroestradiol-(FES) PET/CT, and PET/MRI;
5. ECOG Grade 0 - 2, with minimum life expectancy of at least 3 months;
6. At least one baseline eligible lesion. Per RECIST criteria (version 1.1), an eligible lesion at baseline is considered measurable when ≥ 10mm diameter in the longest diameter;
7. Willing to refrain from using lotions, creams, etc. during the treatment period;
8. Subjects with adequate organ and bone marrow function as defined below:

   * ANC ≥ 1,500/µl
   * Hemoglobin ≥ 9.5 grams/dL
   * Platelets ≥ 75,000/µl
   * AST (aspartate transaminase or SGOT)/ALT (alanine aminotransferase or SGPT) ≤ 3.0 x ULN and total bilirubin ≤ 2.0 x ULN with no evidence of cholestasis
   * Creatinine ≤ 1.5x ULN;
9. Last dose of any systemic non-taxane cytotoxic chemotherapy completed at least one day prior to Day 1. Last dose of any systemic taxane cytotoxic chemotherapy completed at least 4 weeks prior to Day 1
10. Willing to use appropriate birth control for patients of child-bearing potential;
11. Abstinence from all manner of physical contact near the treatment area during and up to 2 weeks after the treatment phase.

Exclusion Criteria:

1. Open or ulcerated wound(s) extending through the dermis within the treatment area;
2. Colorectal, hepatocellular, gallbladder, cholangiocarcinoma, neuroendocrine, melanomas, hematological and central nervous system (CNS) malignancies;
3. Active viral hepatitis A, B, or C or preexisting or acute liver disease;
4. Systemic treatment or localized treatment to target area with the following within the 4 weeks prior to the first treatment visit: radiotherapy, intralesional therapy; laser therapy surgery (other than biopsy), local hyperthermia, levulinic acid, 5-fluorouracil, high potency corticosteroids (including systemic steroids), retinoids, diclofenac, hyaluronic acid, imiquimod;
5. Elective surgery for treatment of the cutaneous metastases during the study and up to 4 weeks after the treatment period. Cutaneous metastases are required to remain in-situ and measurable for up to 2 weeks after last treatment to achieve study objectives;
6. Known allergic reactions, irritations or sensitivity to the active ingredients or other components of SOR007;
7. Symptoms of a clinically significant illness that may place the subject at risk by trial participation or influence the outcome of the trial in the four weeks before first treatment and during the trial;
8. Participation in the treatment phase of another clinical trial within the four weeks prior to treatment in this clinical trial;
9. Investigator's opinion of subject's probable noncompliance or inability to understand the trial and/or give adequate informed consent;
10. Evidence of current chronic alcohol or drug abuse;
11. Pregnancy and/or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Marie Cavanna-Mast, Study Director — US Biotest; Julie E Lang, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacouture ME, Goldfarb SB, Markova A, Chawla SP, Dewnani K, Iacobucci M, Lang JE. Phase 1/2 study of topical submicron particle paclitaxel for cutaneous metastases of breast cancer. Breast Cancer Res Treat. 2022 Jul;194(1):57-64. doi: 10.1007/s10549-022-06584-6. Epub 2022 Apr 26. PMID 35471470

RESULTS

PARTICIPANT FLOW:
Groups:
- SOR007 2.0% Group A: 2.0% SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment applied topically twice daily for 28 days
  SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment: One (1) Finger Tip Unit (FTU), or approximately 0.5 g, of SOR007 ointment will be applied topically to a 50 cm2 treatment area.
- SOR007 2.0% Group B: 2.0% SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment applied topically twice daily for 56 days
  SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment: One (1) Finger Tip Unit (FTU), or approximately 0.5 g, of SOR007 ointment will be applied topically to a 50 cm2 treatment area.
Period: Overall Study
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B
Started | 4 | 3 | 5 | 11
Completed All Dosing | 3 | 3 | 3 | 10
Completed | 1 | 3 | 3 | 5
Not Completed | 3 | 0 | 2 | 6
Not completed — Non-compliance with study schedule | 1 | 0 | 0 | 1
Not completed — Decision to start another clinical trial. Not related to AE. | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Oncologist decision to start subject on IV chemotherapy prohibited under protocol. | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B | Total
Number analyzed (Participants) | 4 | 3 | 5 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (12.7) | 66.3 (8.3) | 63.2 (11.3) | 63.0 (10.8) | 63.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 10 | 21
  Male | 0 | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 1 | 5
  Not Hispanic or Latino | 3 | 2 | 3 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 3
  White | 4 | 3 | 1 | 6 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.23 (4.51) | 26.13 (3.96) | 29.54 (4.94) | 25.05 (5.21) | 25.85 (5.07)
ECOG Performance Status [Mean (Standard Deviation); unit: units on a scale] — The ECOG performance status scale is a measurement that describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. The scale ranges from 0 to 5, with a lower score indicating a more functional patient and a higher score indicating a patient with more negative impacts to their daily functions.
  units on a scale | 1.0 (0.8) | 0.7 (0.6) | 0.6 (0.9) | 0.7 (0.5) | 0.7 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Treatment emergent adverse events will include all reported adverse events, laboratory assessments, physical examination findings, and vital signs.
Time Frame: Baseline through Day 59 (for 28 days of treatment) or Day 86 (for 56 days of treatment)
Population: All subjects who received SOR007 were included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B
Number analyzed (Participants) | 4 | 3 | 5 | 11
Participants | 4 | 3 | 5 | 10

2. Secondary Outcome: Objective Clinical Response
Description: Objective Clinical Response (Complete Clinical Response (CR) + Partial Response (PR)) is defined as the percentage of study subjects who achieve complete clinical response or partial response 14 days after last treatment (Day 43 or Day 70).
  Complete clinical response (CR) is defined as absence of any detectable residual disease in the treatment area; partial response (PR) as at least a 30% decrease in the sum of the diameters of eligible lesion(s) within the treatment area compared to baseline; progressive disease (PD) as at least a 20% increase in the sum of diameters of eligible lesion(s) within the treatment area, taking as reference the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); and stable disease (SD) as between that defined as PR or PD. Eligible lesions will be determined at baseline by the RECIST definition of measurable tumors (≥ 10mm in its longest diameter).
Time Frame: Baseline and Day 43 (for 28 days of treatment) or Day 70 (for 56 days of treatment)
Population: Of the 23 Subjects enrolled, evaluable photography 14 days after the last dose of SOR007 was provided in 14 (60.9%) Subjects; two in the 0.15% treatment group, three in the 1.0% treatment group, four in 2.0% A treatment group, and five in 2.0% B treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B
Number analyzed (Participants) | 2 | 3 | 4 | 5
Participants
  Complete Response | 0 | 0 | 0 | 1
  Partial Response | 0 | 2 | 0 | 0
  Progressive Disease | 1 | 0 | 3 | 0
  Stable Disease | 1 | 1 | 1 | 4

3. Secondary Outcome: Change in Pain at the Treatment Area
Description: Change in pain at the treatment area will be measured by the Numeric Rating Scale (NRS-11). The numerical scale ranges from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable." A lower score equates to less severe pain (better outcome) and a higher score equates to more severe pain (worse outcome).
Time Frame: Baseline and Day 43 (for 28 days of treatment) or Day 70 (for 56 days of treatment)
Population: All subjects who received SOR007 were included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B
Number analyzed (Participants) | 4 | 3 | 5 | 11
units on a scale
  Baseline (Day 1) | 0.0 (0.0) | 0.3 (0.6) | 1.4 (1.3) | 1.1 (2.0)
  2 Weeks after Last Dose (Day 43 for 28-day treatment groups or Day 70 for 56-day treatment groups) | 0.0 (0.0) | 1.0 (1.7) | 3.8 (2.6) | 0.3 (0.7)

4. Secondary Outcome: Objective Tumor Response (OTR)
Description: Objective Tumor Response (OTR), defined as the difference in the lesion size within the treatment area between baseline and 14 days after the last dose in the dose group i.e. Day 43 for dose escalation Subjects, and dose expansion Group A Subjects; Day 70 for dose expansion Group B Subjects; or between baseline and last tumor assessment for early terminators. Four OTRs are calculated based on different definitions of "lesion size": 1) Area of the primary eligible lesion, 2) Sum of area of all eligible lesions, 3) Longest diameter of the primary eligible lesion, and 4) Sum of longest diameter of all eligible lesions.
Time Frame: Baseline and Day 43 (for 28 days of treatment) or Day 70 (for 56 days of treatment)
Population: One subject in SOR007 2.0% Group A was not included in the analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0%
Number analyzed (Participants) | 4 | 3 | 15
mm^2
  Based on Area of the Primary Eligible Lesion | -31.03 (22.00) | 302.63 (330.55) | -165.05 (679.24)
  Based on Total Area of all Eligible Lesions | -40.57 (25.56) | 407.33 (499.66) | -176.61 (883.76)
  Based on Longest Diameter of the Primary Eligible Lesion | -5.50 (9.75) | 5.11 (6.55) | -0.96 (16.57)
  Based on Total Longest Diameter of all Eligible Lesions | -5.75 (9.58) | 4.88 (6.17) | 1.26 (37.34)

ADVERSE EVENTS:
Time Frame: The Investigator recorded all reportable events with start dates occurring any time after first study drug dose application until 30 days after the last study drug application, or in the case of an TESAE, at least 30 days after onset, whichever was later.
Description: AEs were collected at all study visits from the time of first study drug application. Study personnel were required to review the Subject's diary at each visit to confirm it was adequately completed and to address and document discrepancies, missing entries and errors. Study personnel also asked open-ended questions to obtain information about AEs at every visit.
Arm/Group | SOR007 0.15% | SOR007 1.0% | SOR007 2.0% Group A | SOR007 2.0% Group B
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 2/5 | 4/11
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 5/5 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOR007 0.15% (N=4) | SOR007 1.0% (N=3) | SOR007 2.0% Group A (N=5) | SOR007 2.0% Group B (N=11)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOR007 0.15% (N=4) | SOR007 1.0% (N=3) | SOR007 2.0% Group A (N=5) | SOR007 2.0% Group B (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Application site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pain (General disorders) | 1 (1) | 1 (1) | 2 (7) | 3 (4)
Application site pruritus (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Application site wound (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site haemorrhage (General disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Crepitations (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corynebacterium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Facial wasting (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT03101358/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT03101358/SAP_001.pdf